CLINICAL TRIAL: NCT02864875
Title: Early Administration of Fibrinogen Concentrate in Polytraumatized Patients With Thromboelastometry Suggestive of Hypofibrinogenemia: a Randomized Feasibility Trial
Brief Title: Early Administration of Fibrinogen in Polytraumatized Patients With Hypofibrinogenemia: a Randomized Feasibility Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Lucas Siqueira de Lucema, Lucas Lucena, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 662.182
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Trauma; Bleeding Disorder; Fibrinogen; Deficiency, Acquired
Keywords: Trauma; Coagulopathy; Fibrinogen; Fibrinogen Concentrate; Thromboelastometry; Hypofibrinogenemia; Early Fibrinogen Replacement
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders; Afibrinogenemia | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Not to receive an early replacement of fibrinogen
- Intervention (Experimental): Receive early replacement through fibrinogen concentrate (50mg per kg of body weight)
  Interventions: Drug: Fibrinogen concentrate

INTERVENTIONS:
Drug: Fibrinogen concentrate — Receive fibrinogen concentrate 50mg/kg of body weight after randomization
  Other Names: Haemocomplettan®
  Arms: Intervention

SUMMARY:
This is a randomized feasibility trial conducted with severe trauma patients. At admission patients presented hypofibrinogenemia, hypotension and tachycardia. The primary outcome was feasibility assessed by the proportion of patients receiving the allocated treatment up to 60 minutes after randomization. The treatments regards to receive or not to receive an early replacement of fibrinogen.

DETAILED DESCRIPTION:
This is a randomized feasibility trial conducted between December 2015 and January 2017 with severe trauma patients (Index of Shock Severity [ISS] ≥ 15) admitted to the emergency room of a large trauma center. At admission patients presented qualitative hypofibrinogenemia (FIBTEM A5 ≤ 9 mm), hypotension (systolic blood pressure <90 mmHg) and tachycardia (heart rate > 100 bpm). The primary outcome was feasibility assessed by the proportion of patients receiving the allocated treatment up to 60 minutes after randomization meaning receive replacement through fibrinogen concentrate (50mg per kg of body weight) by the intervention group and not to receive an early replacement of fibrinogen by control group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Severe trauma patients (Index of Shock Severity [ISS] ≥ 15)
* Hypotension (systolic blood pressure < 90 mmHg)
* Tachycardia (heart rate > 100 bpm)
* Qualitative hypofibrinogenemia (FIBTEM A5 ≤ 9 mm)

Exclusion Criteria:

* Patient or family do not agree to sign the informed consent form
* Eligible for institutional massive transfusion protocol
* Pregnant
* Previous coagulopathy disorders
* Use of anticoagulants drugs and/or platelet anti aggregation drugs (exception for aspirin)
* Previous thromboembolic disorders or events
* Cardiopulmonary arrest before hospital admission
* Patient admitted after another hospital transfer
* Time from trauma to screening above six hours
* Patients with exclusively traumatic brain injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by the proportion of patients receiving the allocated treatment up to 60 minutes after randomization | 60 minutes
  The proportion of patients receiving the allocated treatment up to 60 minutes after randomization

SECONDARY OUTCOMES:
Overall blood tube drainage | 48 hours
  Overall blood tube drainage
Overall blood tube drainage | Up to four weeks - Through the length of hospital stay
  Overall blood tube drainage
Transfusion requirements assessed as units of red blood cell, fresh frozen plasma, blood platelets and cryoprecipitate | 48 hours
  Transfusion requirements
Transfusion requirements assessed as units of red blood cell, fresh frozen plasma, blood platelets and cryoprecipitate | Up to four days - Through the Length of operating room stay
  Transfusion requirements
Transfusion requirements assessed as units of red blood cell, fresh frozen plasma, blood platelets and cryoprecipitate | Up to four weeks - Through the Length of intensive care unit stay
  Transfusion requirements
Transfusion requirements assessed as units of red blood cell, fresh frozen plasma, blood platelets and cryoprecipitate | Up to four weeks - Through the Length of operating room stay
  Transfusion requirements
Costs of blood therapy assessed by de median value spent on each patient due to red blood cell, fresh frozen plasma, blood platelets, cryoprecipitate and fibrinogen concentrate | Up to four weeks - Through the Length of operating room stay
  Costs of blood therapy
Thromboembolic events assessed by any clinical manifestation that can be related to a thromboembolic event | First two weeks after hospital admission
  Thromboembolic events
Reoperate due to bleeding | Up to four weeks - Through the Length of operating room stay
  Reoperate due to bleeding
Ventilator-free days | Up to four weeks - Through the Length of operating room stay
  Ventilator-free days
Vasopressor-free days | Up to four weeks - Through the Length of operating room stay
  Vasopressor-free days
Length of hospital stay | Up to four weeks - Through the Length of operating room stay
  Length of hospital stay
Length of intensive care unit stay | Up to four weeks - Through the Length of intensive care unit stay
  Length of intensive care unit stay
In-hospital Deaths | Up to four weeks - Through the Length of operating room stay
  In-hospital Deaths
Sequential Organ Failure Assessment (SOFA) score on the first day after intensive care unit admission | First day after intensive care unit admission
  The Sequential Organ Failure Assessment (SOFA) score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems.
  The SOFA score can be used to determine the level of organ dysfunction and the mortality risk in ICU patients.
  High values means worst outcomes
Sequential Organ Failure Assessment (SOFA) score on the fifth day after intensive care unit admission | Fifth day after intensive care unit admission
  The Sequential Organ Failure Assessment (SOFA) score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems.
  The SOFA score can be used to determine the level of organ dysfunction and the mortality risk in ICU patients.
  High values means worst outcomes
Sequential Organ Failure Assessment (SOFA) score on the seventh day after intensive care unit admission | Seventh day after intensive care unit admission
  The Sequential Organ Failure Assessment (SOFA) score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems.
  The SOFA score can be used to determine the level of organ dysfunction and the mortality risk in ICU patients.
  High values means worst outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Lucas S Lucena, MD, Principal Investigator — Hospital das Clínicas da FMUSP
Locations (1):
- Hospital das Clínicas - FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucena LS, Rodrigues RDR, Carmona MJC, Noronha FJD, Oliveira HP, Lima NM, Pinheiro RB, Silva WAD, Cavalcanti AB. Early administration of fibrinogen concentrate in patients with polytrauma with thromboelastometry suggestive of hypofibrinogenemia: A randomized feasibility trial. Clinics (Sao Paulo). 2021 Nov 8;76:e3168. doi: 10.6061/clinics/2021/e3168. eCollection 2021. PMID 34755760